CLINICAL TRIAL: NCT04882566
Title: Assessment of Nutritional Knowledge in Patients With Inflammatory Bowel Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Kerollos Latif Labib, Principle investigator of Internal Medicine department, Assiut University
Other Study IDs: Nutrition in IBD patients
Record Dates: First submitted 2021-03-17; First posted 2021-05-12 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Ulcerative Colitis; Crohn Disease; Nutrition
Keywords: Paleolithic; Nutrition; Questionnaire; Inflammatory Bowel Disease; Nutritional assessment; Ulcerative colitis; Crohn's disease; Diet
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease; Inflammatory Bowel Diseases | interventions — Diet, Paleolithic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Paleolithic Diet — Advice to follow Paleolithic Diet for Inflammatory bowel disease Patients

SUMMARY:
Patients with inflammatory bowel disease (IBD) are increasingly becoming interested in nonpharmacologic approaches to their disease. One of the most frequently asked questions of IBD patients is what they should eat. The role of diet has become very important in the prevention and treatment of IBD. Although there is a general lack of rigorous scientific evidence that demonstrates which diet is best for certain patients, several diets have become popular.

Aim of the Work To assess IBD patients' knowledge about the role of nutrition in the management of their Inflammatory Bowel Disease and the dietary beliefs, behaviors, and daily dietary practices in adult IBD patients that they make to avoid exacerbation of disease symptoms or to gain more control of bowel symptoms, keeping in mind our traditional and oriental food and food habits in Egypt.

Also to evaluate the role of one of the most common dietary regimens; the Paleolithic diet in active mild or moderate inflammatory bowel disease.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD) is a chronic auto-immune disorder with unclear etiology. Multiple factors play a role in the patho¬genesis of IBD. These may include diet, environmental factors, immunologic factors, infectious agents, genetic susceptibility, and the microbiome. The emergence of rapid increases in the incidence of IBD over the past several decades in low-incidence parts of the world, clearly points to the important role that the environment plays in disease develop¬ment.

In Egypt, it was noticed a marked increase in the frequency of both UC and CD diagnoses during the most recent 10 years from 1995 to 2009 and it is still rising till now .

Therefore, clinicians, along with patients, have questioned whether diet influences the onset, prognosis, and the need of drug intensification ( Figure 2 ). The ques¬tion of what to eat is the most commonly encountered question as well as the most challenging one asked to gastroenterologists managing IBD patients. At present, there is no specific IBD diet that is supported by robust data, leaving patients to seek nonmedical resources for dietary advice. Dietary intervention trials have been limited by their lack of a placebo control group and the difficulty in meticulously capturing dietary intake conjointly with the potential for complex interactions between foods. Furthermore, dietary trials may not detect significant dif¬ferences for patients undergoing withdrawal of specific drug therapies.

The lay literature has promoted several popular diets that have been touted to alleviate intestinal inflammation and have thereby been advocated for patients with IBD. These include the specific carbohydrate diet (SCD); the low-fermentable oligosaccharide, disaccharide, monosaccharide, and polyol (Low-FODMAP) diet; the Paleolithic diet (Paleo); and the anti-inflamma¬tory diet (IBD-AID). As patients look to complementary therapies for the management of their disease, clinicians must understand the effectiveness and the role of these dietary interventions to advise and direct patients So that it's clear that access to proper dietary guidance is an essential part of dietary self-management in IBD.However, patients learn about their food tolerances and intolerances by trial and error rather than under the guidance of a health professional. This creates the risk of (micro) nutrient deficiencies in the case of uninformed or badly informed food avoidance and strict diets. Moreover, there is no guarantee that the best possible measures are taken to control the bowel disorder. There is, however, evidence that the effectiveness of personal diets could be improved by the guidance of a professional dietary IBD service.

As a start, it is important to learn more about the current practices and beliefs of IBD patients concerning their diet.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed to have Inflammatory bowel disease either Crohn's disease or Ulcerative Colitis attending our Inflammatory bowel disease outpatient clinic at Al-Rajhy Liver Hospital for any reason, either in remission or in activity at Al-Rajhy Liver Hospital at Al-Rajhy Liver Hospital were included in our study.

Exclusion Criteria:

* Severe disease and critical patients in the Intensive Care Unit with severe exacerbation were excluded from the study. Patients who were not surely diagnosed to have IBD were excluded from the study. Patients with pure perianal CD, a current stoma, previous extensive GI resection, or a current stricture were excluded. Patients were excluded if they had significant comorbidities, or if they were pregnant or lactating. Also, patients with any other acute illness and those who underwent gastrointestinal surgical interventions due to any cause were excluded from the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with Inflammatory Bowel disease either Ulcerative colitis or Crohn's disease who are in remission and activity.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Evaluation of nutritional knowledge among IBD patients | 1 year
  A self-administered questionnaire was formed of 30 questions assessing the following sub-domains. The questionnaire was developed after reviewing the literature on IBD patient's dietary habits, beliefs, therapies, and attitudes. Based on this literature study, relevant topics for the questionnaire were identified. Also, the draft questionnaire was thoroughly discussed with the IBD patient and modified because of practical aspects and face validity. The questionnaire included 30 close-ended questions, which were divided into 5 sub-domains:
  1. General characteristics of the participants ( age, sex, residency, occupation, special habits, IBD type, IBD site in the GIT, disease activity, type of medication, and if there were any complications)
  2. Nutritional knowledge
  3. Dietary beliefs
  4. Dietary behaviors and practices
  5. The source of the dietary advice.

OTHER OUTCOMES:
Role of Paleolithic diet in improving IBD patients symptoms | 1month
  Scientific-based dietary advice with the Paleolithic diet was given to patients who have mild to moderately active disease. Evaluation of the effect of diet in improving IBD patients symptoms is measured using recent standardized and validated questionnaires such as the irritable bowel severity scoring system (IBS-SSS) for evaluation of disease symptoms
  The (IBS-SSS) maximum achievable score is 500 means the worst condition
Role of Paleolithic diet in improving IBD patients Quality of Life | 1 month
  Scientific-based dietary advice with the Paleolithic diet was given to patients who have mild to moderately active disease. Evaluation of the effect of diet in improving IBD patients Quality of Life . We will use the validated Crohn's and ulcerative colitis questionnaire-8 (CUCQ-8) to assess the change in the quality of life before and after the diet trial.
  The (CUCQ-8) maximum achievable score is 700 means the worst condition .
Role of Paleolithic diet in induction of laboratory Remission by its effect on CRP | 1 month
  Also we will assess the serum inflammatory markers such as C-reactive protein (CRP) before and after the diet trial.CRP is measured in milligrams per Liter.
Role of Paleolithic diet in induction of laboratory Remission by its effect on ESR | 1 month
  we will assess the serum inflammatory markers such as Erythrocyte sedemintation rate (ESR) before and after the diet trial. ESR is measured in millimeter per hour.

CONTACTS AND LOCATIONS:
Overall Officials: Kerollos L Labib, MSC, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Knight-Sepulveda K, Kais S, Santaolalla R, Abreu MT. Diet and Inflammatory Bowel Disease. Gastroenterol Hepatol (N Y). 2015 Aug;11(8):511-20. PMID 27118948
- [Background] Lee D, Albenberg L, Compher C, Baldassano R, Piccoli D, Lewis JD, Wu GD. Diet in the pathogenesis and treatment of inflammatory bowel diseases. Gastroenterology. 2015 May;148(6):1087-106. doi: 10.1053/j.gastro.2015.01.007. Epub 2015 Jan 15. PMID 25597840
- [Background] Esmat S, El Nady M, Elfekki M, Elsherif Y, Naga M. Epidemiological and clinical characteristics of inflammatory bowel diseases in Cairo, Egypt. World J Gastroenterol. 2014 Jan 21;20(3):814-21. doi: 10.3748/wjg.v20.i3.814. PMID 24574754